CLINICAL TRIAL: NCT04456803
Title: A Study to Evaluate the Efficacy and Safety of Ferric Citrate Tablet for the Treatment of Hyperphosphatemia in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Brief Title: Ferric Citrate for the Treatment of Hyperphosphatemia in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinomune Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS-CO-1642; CTR20190978 (Other: http://www.chinadrugtrials.org.cn/)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hyperphosphatemia; End Stage Renal Disease; ESRD
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — ferric citrate; Sevelamer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric citrate tablet (Experimental): Ferric citrate arm will receive ferric citrate tablets three times a day with each meal.
  Interventions: Drug: Ferric citrate tablet
- Sevelamer carbonate tablet (Active Comparator): Sevelamer carbonate arm will receive sevelamer carbonate tablets three times a day with each meal.
  Interventions: Drug: Sevelamer carbonate tablet

INTERVENTIONS:
Drug: Ferric citrate tablet — 250mg/tablet, manufactured by Sinomune Pharmaceutical
  Arms: Ferric citrate tablet
Drug: Sevelamer carbonate tablet — 800 mg/tablet, manufactured by Genzyme Ireland Limited
  Other Names: Renvela
  Arms: Sevelamer carbonate tablet

SUMMARY:
To evaluate the efficacy and safety of ferric citrate tablet in the control of serum phosphorus levels in patients with chronic kidney disease undergoing hemodialysis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, parallel, phase III study. This study is consisting of a Screening/Washout period (14 days) and a Treatment/Observation period (12 weeks). The subjects with regular hemodialysis should stop using the phosphorus binder before the Washout period. During the Treatment period, the subjects will be randomly assigned to the ferric citrate tablets group (study group) or sevelamer carbonate tablet group (control group) in the ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 18 and 75 years (including the boundary value) and no gender limitation;
2. Patients who maintain the hemodialysis schedule (including hemofiltration (HF) hemodialysis (HDF) hemoperfusion (HP)) as not less than 3 times a week in the 3 months before random enrollment.
3. Patients with a serum phosphorus level between 1.97 to 3.23 mmol/L (excluding the boundary value) after washout.
4. Kt/Vurea ≥1.2 or URR ≥65%.
5. Before the screening period, CKD-MBD related drug treatment is stable for more than one month, including the use of vitamin D (active vitamin D, vitamin D analogues, etc.) or calcimimetics (cinacalcet, etc.) and the dose remains unchanged.
6. The expected survival is greater than 6 months.
7. Willing to give written informed consent.

Exclusion Criteria:

1. Patients with a serum ferritin level ≥800 ng/mL or TSAT ≥50%.
2. Patients with hemochromatosis or patients receiving treatment for iron overload, or patients with paroxysmal sleep hemoglobinuria.
3. Patients who received blood transfusions within 3 months prior to Screening, or patients with hemoglobin ≤60 g/L.
4. Patients with intact-PTH >1000 pg/mL
5. Patients complicated with any of the following gastrointestinal diseases: acute peptic ulcer, chronic ulcerative colitis, localized enteritis, intestinal obstruction, habitual constipation (number of stools once per week), and chronic diarrhea (number of stools four times per day), or patients with a history of gastrectomy or enterectomy or patients who had undergone gastrointestinal surgery within 3 months prior to Screening, or patients with dysphagia.
6. Patients with impaired liver function (hepatic dysfunction or serum total bilirubin, aspartate aminotransferase or alanine aminotransferase ≥ 2 times the upper limit of normal) or patients with cirrhosis.
7. Patients with a history of parathyroidectomy (PTx) or percutaneous anhydrous ethanol injection (PEIT) within 6 months.
8. Patients with uncontrolled diabetes or uncontrolled high blood pressure or current active infectious diseases such as active viral hepatitis.
9. Patients with a history of severe allergies may be allergic to research drugs.
10. Patients with cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.) or cardiovascular disease (congestive heart failure of Class III or severer in NYHA classification) requiring hospitalization within 6 months prior to Screening, or patients who use antiarrhythmic drugs to control arrhythmias or who use antiepileptic drugs to control seizures.
11. Patients who plan to receive a kidney transplant during the study period.
12. Patients with a history of drug and alcohol abuse
13. Patients with active or advanced malignancy.
14. Women who are pregnant or lactating
15. Patients complicated with active bleeding or requiring anticoagulation therapy with citrate in hemodialysis
16. Patients who had participated in other clinical studies within 1 month prior to Screening.
17. Patients who are not suitable for participating in the trial according to the investigator's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
The change in serum phosphorus levels | 12 Weeks
  The change in serum phosphorus levels at the end of treatment as compared to baseline (before the first dose).

SECONDARY OUTCOMES:
Changes in serum phosphorus levels | week 2, 4, 6, 8
  Changes in serum phosphorus levels from baseline
Area under the curve of serum phosphorus level | week 0, 2, 4, 6, 8, 12
  Area under the curve of serum phosphorus level to visit time (AUC 0-12 weeks)
The proportion of subjects whose serum phosphorus levels reached the target | week 4, 6, 8 and 12
  The proportion of subjects whose serum phosphorus levels reached the target range at week 4, 6, 8 and 12 of treatment (the standard was defined as blood phosphorus ≤1.78mmol /L, and ≥1.13mmol /L).
The change in serum calcium (corrected) levels. | week 4, 8 and 12
  The change in serum calcium (corrected) levels at week 4, 8 and 12 of treatment as compared to baseline.
The change in the level of intact-PTH levels. | week 4, 8 and 12
  The change in the level of intact-PTH levels at week 4, 8 and 12 of treatment as compared to baseline.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - The first affiliated hospital of Baotou medical college, Baotou
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - The second hospital of Dalian medical university, Dalian
  - The affiliated hospital of Inner Mongolia Medical University, Hohhot
  - The second people's hospital of Huaian, Huai'an
  - Jinan central hospital, Jinan
  - Shandong province Qianfoshan hospital, Jinan
  - Zhongnan Hospital Southeast University, Nanjing
  - The people's hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Shenzhen people's hospital, Shenzhen
  - The third hospital of Hebei medical university, Shijiazhuang
  - General Hospital of Tianjin Medical University, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan provincal people's hospital, Zhengzhou
  - Zhengzhou People's Hospital, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou